CLINICAL TRIAL: NCT04208802
Title: Effect of Smoking on Saliva Composition and the Development of Dental Erosion - an In-situ Study
Brief Title: Effect of Smoking on Saliva Composition and the Development of Dental Erosion
Status: Completed | Type: Observational
Sponsor: University of Göttingen (Other)
Responsible Party: Principal Investigator, Philipp Kanzow, Prof. Dr. med. dent., Dr. rer. medic., Senior Dental Practitioner, University Medical Center Goettingen
Other Study IDs: Erosion-Smoking; 15/10/19 (Other: Local Ethics Commission); 02785 (Other: UMG study center)
Record Dates: First submitted 2019-12-18; First posted 2019-12-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Dental Erosion
MeSH Terms: conditions — Tooth Erosion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples are obtained and retained for 10 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Smokers: Volunteers smoking at least 10 cigarettes per day
  Interventions: Other: Use of fluoridated toothpaste; Other: Wearing of an intraoral device with bovine tooth samples; Other: Wearing of an intraoral device with resin samples
- Non-smokers: Non-smoking volunteers
  Interventions: Other: Use of fluoridated toothpaste; Other: Wearing of an intraoral device with bovine tooth samples; Other: Wearing of an intraoral device with resin samples

INTERVENTIONS:
Other: Use of fluoridated toothpaste — Use of fluoridated toothpaste
Other: Wearing of an intraoral device with bovine tooth samples — Wearing of an intraoral device with bovine tooth samples
Other: Wearing of an intraoral device with resin samples — Wearing of an intraoral device with resin samples

SUMMARY:
The aim of this study is to investigate whether smoking is associated with changes in salivary composition and/or predisposition to erosion.

Healthy volunteers are observationally wearing an intraoral device with both bovine tooth specimens (enamel and dentin) and resin specimens twice for two hours each. Afterwards, specimens are eroded extraorally and calcium release into the acid is measured.

Total protein concentration and protein composition of the salivary pellicles on the resin samples are measured. Additionally, salivary parameters (unstimulated and stimulated saliva flow rate, pH, buffer capacity, total protein content and protein composition as well as concentration of inorganic calcium, phosphate, and fluoride) are measured.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers aged between 20 and 50 years who are able to give written consent

Exclusion Criteria:

* Non-fulfillment of the inclusion criteria
* Intake of medications or diseases altering salivary secretion
* Refusal to use fluoridated toothpastes
* Known allergies to substances used in the study
* Orthodontic treatment or malfunction which does not allow wearing an intraoral device

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Exploratory study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Calcium release from bovine enamel and dentin specimens by extraoral erosion (nmol/Square Millimeter). | Immediately after the intraoral device has been worn once for two hours.

SECONDARY OUTCOMES:
Determination of unstimulated and stimulated saliva flow rate (mL/min). | Saliva samples are collected for 5 min each on three visits.
Determination of saliva pH (pH). | Saliva samples are collected for 5 min each on three visits.
Determination of salivary buffer capacity (pH). | Saliva samples are collected for 5 min each on three visits.
Determination of total protein content (mg/L) and protein composition (qualitatively) in saliva. | Saliva samples are collected for 5 min each on three visits.
Determination of inorganic calcium (mmol/L), phosphate (mmol/L) and fluoride (µmol/L) in saliva. | Saliva samples are collected for 5 min each on three visits.
Determination of total protein concentration (ng/Square Millimeter) and protein composition (qualitatively) within the salivary pellicles. | Immediately after the intraoral device with resin samples has been worn once for two hours.

CONTACTS AND LOCATIONS:
Overall Officials: Annette Wiegand, Prof. Dr. med. dent., Principal Investigator — Dept. of Prev. Dentistry, Periodontology and Cariology, University Medical Center Göttingen, Germany
Locations (1):
- University Medical Center Göttingen, Dept. of Preventive Dentistry, Periodontology and Cariology, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carpenter G, Cotroneo E, Moazzez R, Rojas-Serrano M, Donaldson N, Austin R, Zaidel L, Bartlett D, Proctor G. Composition of enamel pellicle from dental erosion patients. Caries Res. 2014;48(5):361-7. doi: 10.1159/000356973. Epub 2014 Mar 6. PMID 24603346
- [Background] Moazzez R, Bartlett D. Intrinsic causes of erosion. Monogr Oral Sci. 2014;25:180-96. doi: 10.1159/000360369. Epub 2014 Jun 26. PMID 24993266
- [Background] Wiegand A, Bliggenstorfer S, Magalhaes AC, Sener B, Attin T. Impact of the in situ formed salivary pellicle on enamel and dentine erosion induced by different acids. Acta Odontol Scand. 2008 Aug;66(4):225-30. doi: 10.1080/00016350802183401. PMID 18607835
- [Background] Wiegand A, Meier W, Sutter E, Magalhaes AC, Becker K, Roos M, Attin T. Protective effect of different tetrafluorides on erosion of pellicle-free and pellicle-covered enamel and dentine. Caries Res. 2008;42(4):247-54. doi: 10.1159/000135669. Epub 2008 Jun 4. PMID 18523383
- [Background] Zwier N, Huysmans MC, Jager DH, Ruben J, Bronkhorst EM, Truin GJ. Saliva parameters and erosive wear in adolescents. Caries Res. 2013;47(6):548-52. doi: 10.1159/000350361. Epub 2013 Jun 15. PMID 23774653
- [Background] Kanzow P, Wegehaupt FJ, Attin T, Wiegand A. Etiology and pathogenesis of dental erosion. Quintessence Int. 2016 Apr;47(4):275-8. doi: 10.3290/j.qi.a35625. PMID 27022647
- [Background] Wiegand A, Rosemann A, Hoch M, Barke S, Dakna M, Kanzow P. Erosion-Protective Capacity of the Salivary Pellicle of Female and Male Subjects Is Not Different. Caries Res. 2019;53(6):636-642. doi: 10.1159/000500046. Epub 2019 Jun 4. PMID 31163440
- [Result] Kanzow P, Lenz C, Schlarmann F, Barke S, Rohland B, Schmidt A, Gorshkova A, Neuenroth L, Wiegand A. Saliva and salivary pellicle composition and proteomic profile in smokers vs. non-smokers and its effect on dental erosion. J Dent. 2026 Jan 21:106517. doi: 10.1016/j.jdent.2026.106517. Online ahead of print. PMID 41577165